CLINICAL TRIAL: NCT06038695
Title: Ultrasound-based Imaging to Detect Early Changes of Hard and Soft Tissue Around Immediately Placed Implants With Volume-Stable Collagen Matrix Combined With rhPDGF-BB: Pilot Study
Brief Title: Immediate Implant Placement Using Volume-Stable Collagen Matrix Combined With rhPDGF-BB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Currently, there is no capacity for this project in the institute
Sponsor: I-Ching Wang (Other)
Responsible Party: Sponsor-Investigator, I-Ching Wang, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202212227
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Tooth Extraction; Immediate Implant Placement
MeSH Terms: interventions — Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Xenogeneic Volume-Stable Collagen (VCMX) graft with growth factor-BB (Experimental): Subjects in this arm will have a xenogeneic volume-stable collagen matrix in combination with recombinant human platelet-derived growth factor-BB at the time of immediate implant placement.
  Interventions: Device: Xenogeneic Volume-Stable Collagen (VCMX) graft with growth factor-BB

INTERVENTIONS:
Device: Xenogeneic Volume-Stable Collagen (VCMX) graft with growth factor-BB — * Fibro-Gide is the Volume-Stable Collagen Matrix.
  * Recombinant human platelet-derived growth factor-BB will be found within the device of GEM21S.
  Other Names: Fibro-Gide, Geistlich Pharma; GEM21S, Lynch Biologics

SUMMARY:
The goal of this study is to test a volume-stable collagen matrix in combination with recombinant human platelet-derived growth factor-BB, specifically in patients who have an immediate implant placement for teeth #5-#12.

The main question this study aims to answer is does the recombinant human platelet-derived growth factor-BB accelerate the formation of blood vessels and augment tissue volume around the immediate implant.

Participants will be asked to undergo immediate implant placement using volume-stable collagen matrix in combination with recombinant human platelet-derived growth factor-BB, as well as attend 11 study visits over the course of 1.25 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-95
* Has a single hopeless tooth in the maxillary esthetic zone (i.e., first premolar to first premolar, tooth #5-tooth #13)
* Adequate oral hygiene (i.e., full-mouth bleeding score (FMBS) and full mouth plaque score (FMPS) of less than 25%)
* Adequate tooth space to support an immediate implant placement (i.e., adequate mesiodistal space of greater than or equal to 6 mm and interocclusal space to support a non-occluding provisionalization).
* Postextraction vertical bone defect of the buccal socket wall was less than or equal to 3mm

Exclusion Criteria:

* patients taking long-term (more than 3 months) medications affecting bone metabolism
* generalized untreated periodontitis with greater than of 30% of sites with greater than 5mm pocket depths and bleeding upon probing with a dental probe
* medical contraindications for having a surgical procedure (i.e., ASA Status of III, patient with a severe systemic disease that is not life-threatening; ASA Status of IV, a patient with a severe systemic disease that is a constant threat to life).
* history of radiotherapy in the head and neck region
* heavy smoker (greater than 10 cigarettes per day)
* pregnancy
* gingival recession before extraction in relation to the contralateral tooth

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in from Baseline in Soft and Hard Tissue Thickness as assessed by ultrasound. | Multiple time points (i.e. 0, Immediately after implant placement, 1 week, 2 weeks, 4 weeks, 6 weeks, 12 weeks, 16 weeks, 24 weeks, and 48 weeks after immediate implant placement
  Tissues will be measured in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: I-Ching Wang, DDS,MS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa College of Dentistry and Dental Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No